CLINICAL TRIAL: NCT01820767
Title: Paricalcitol Action on Parameters of Inflammation and Oxidative Stress in Patients With Chronic Kidney Disease Stage Vd Carriers Tunneled Hemodialysis Catheters
Brief Title: Paricalcitol Over Inflammatory Parameters on Chronical Kidney Disease Patients
Acronym: SENPARIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ricardo Mouzo Mirco (Other)
Responsible Party: Sponsor-Investigator, Ricardo Mouzo Mirco, MD, Hospital El Bierzo
Organization: Hospital El Bierzo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SENPARIC-2011-01; NCT02210533 (obsolete NCT alias)
Record Dates: First submitted 2013-03-19; First posted 2013-03-29 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Vd-stadium.; Inflammatory patterns; Paricalcitol; Atorvastatin
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol; Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paricalcitol (Experimental): SUBGROUP 1 (G1): Paricalcitol oral dosis triphosphoinositide mgc/100, 3 days a week.
  Interventions: Drug: Paricalcitol
- Paricalcitol, Atorvastatin (Active Comparator): SUBGROUP 2 (G2): Paricalcitol (same dosis than G1) + Atorvastatin (1 daily dosis 20 mg)
  Interventions: Drug: Paricalcitol, atorvastatin
- Atorvastatin (Active Comparator): SUBGROUP 3 (G3): Atorvastatin (same G2 dosis)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Paricalcitol — Oral Paricalcitol. parathyroid hormone i mcg/100. 3 days per week, the same day as haemodialysis is done, during 12 weeks.
  Other Names: Group 1
  Arms: Paricalcitol
Drug: Paricalcitol, atorvastatin — Oral Paricalcitol. parathyroid hormone i mgc/100. 3 days a week, the same day as haemodialysis, during 12 weeks.
  Atorvastatin: 20 mg/day oral (1 take) during 12 weeks.
  Other Names: G2
  Arms: Paricalcitol, Atorvastatin
Drug: Atorvastatin — Atorvastatin: 20 mg/day oral (1 take) during 12 weeks
  Other Names: G3
  Arms: Atorvastatin

SUMMARY:
Use of Paricalcitol in stage Vd Chronic Kidney Disease patients, over the effect of inflammatory and oxidative stress parameters.

DETAILED DESCRIPTION:
Use of Paricalcitol in stage Vd Chronic Kidney Disease patients using a permanent catheter due to haemodialysis; over the effect of inflammatory and oxidative stress parameters. This study uses paricalcitol (vitamin D) versus atorvastatin versus paricalcitol plus atorvastatin treatments.

ELIGIBILITY:
Inclusion Criteria:

* Vd CKD patients using haemodialysis during 3 or more months.
* Tunnelized-bearer permanent catheters on haemodialysis at last 6 months previous at the beginning of the study. .
* Kt stable, over 45 litres on both sexs.
* Patients in treatment wiht atorvastatin
* Patients without infectious or inflammatory processes over 8 weeks.
* Two consecutive PTH < than 400 pg/ml; Ca<10.2 and P <7.0 mg/dl.

Exclusion Criteria:

* Patients > 18 years.
* Pregnant women.
* Patients hospitalized 4 weeks before the beginning of the treatment.
* Immunosuppressor intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Oxidative stress and inflammative parameters in patients wiht CKD stage Vitamin D after 12 weeks of treatment | 12 weeks of treatment wiht visits and analysis
  Measure parameter: IL-2
Oxidative stress and inflammative parameters | 12 weeks of treatment
  Measure unit: IL-4
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  IL-5
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  IL-6
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  IL-10
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  IL-13
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  TNF-beta
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD3
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD4
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD8
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD19
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD25
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD56
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD69
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  CD95
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  COX-2
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  iNOS
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  PGE2
Oxidative stress and inflammative parameters in patients with CKD stage vitamin D after 12 weeks of treatment | 12 weeks of treatment with visits and analysis
  FGF-23

SECONDARY OUTCOMES:
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Weight
Erythropoietin requirements variations | 12 weeks of treatment with visits and analysis
  Fe
Assess potential benefits inflammatory markers | 12 weeks of treatment with visits and analysis
  PTHi
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Height
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Body Mass Index (BMI)
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Abdominal circumference
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Triceps skin fold circumference
Nutritional Parameters | 12 weeks of treatment with visits and analysis
  Bioimpedance
Anaemia parameters | 12 weeks of treatment
  Hemogram
Anaemia Parameters | 12 weeks of treatment
  Biochemistry
Erythropoietin requirement variations | 12 weeks of treatment with visits and analysis
  Ferritin
Erythropoietin requirement variations | 12 weeks of treatment with visits and analysis
  Transferrin saturation index
Erythropoietin requirements variations | 12 weeks of treatment with visits and analysis
  B12
Erythropoietin requirements variations | 12 weeks of treatment with visits and analysis
  Folic Acid
Assess potential benefits in inflammatory markers | 16 weeks, the complete duration of the study
  Kt

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Mouzo Mirco, MD, Principal Investigator — Hospital El Bierzo, Fuentesnuevas Ponferrada
Locations (2):
- Spain (2):
  - Hospital El Bierzo. Servicio de Nefrología., Ponferrada, (León).
  - Hospital de León, León